CLINICAL TRIAL: NCT05446285
Title: Multiple Sclerosis Outcome Determination Evaluating Real Differences After TimE
Acronym: MODERATE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 16/WS/0017
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated: Patients initiating disease modifying treatment within the first year of diagnosis
  Interventions: Other: Clinical assessment
- Untreated: Patients who do not initiate disease modifying treatment within the first year of diagnosis
  Interventions: Other: Clinical assessment

INTERVENTIONS:
Other: Clinical assessment — All participants will be invited to attend their local research facility to undergo a physical and questionnaire assessment as well as an MRI. Assessments include: Expanded Disability Status Scale, 9-Hole Peg Test, MRI scan, Patient Reported Outcome Measures (MSIS-29, neuroQOL and PROMIS), Brief International Cognitive Assessment for MS)

SUMMARY:
To provide real world evidence evaluating whether a strategy of early initiation and escalation of disease modifying treatment (DMT) in relapsing-remitting multiple sclerosis (RRMS) affects disease outcome over a 10 year period. Our aim is to provide evidence for clinicians and patients regarding the benefits and risks of early initiation and active escalation of disease modifying treatments (DMTs) in relapsing-remitting multiple sclerosis (RRMS), using real world data.

DETAILED DESCRIPTION:
We will compare efficacy and safety outcomes for patients with RRMS managed with a) an early initiation and escalation policy and b) an expectant and delayed treatment policy, using patients from the National Health Service Greater Glasgow and Grampian MS centres. Initiation and escalation of DMTs will be the interventions under study and a detailed contemporary clinico-radiological assessment will be undertaken to compare outcomes in the differently treated cohorts over the first 10 years following diagnosis.

To capture and analyse both prospective and retrospective data we will use the OPTIMISE portal. This is a database tool under development in Imperial College London which aims to provide a secure IT framework to capture patient-centred data in MS research. Its aim is to facilitate the capture of prospective longitudinal, standardised clinical and patient-centred data, ideally with an ease that would allow it to be used as an adjunct to routine clinical practice. It will ultimately provide open-source software for management of MS data, integrating anonymised information from multiple centres. Our proposed registry study will utilise the OPTIMISE portal and platform for data capture and analysis - this will serve to pilot the platform before its implementation on a wider scale in a variety of different projects, including the nationwide Scottish DMT database currently under development.

In order to compare these non-randomised patient groups we will use propensity score matching (PSM). This statistical method can account for all the known variables that inform the decision-making process of DMT initiation and escalation, and is used in observational studies to mimic the process of randomisation. The decision to initiate or escalate DMTs in RRMS in clinical practice is based on both patient and disease related factors. Patients with more clinically severe disease are more likely to have DMTs initiated or escalated. For DMT initiation, we will calculate the propensity score based on known prognostic factors at the time of diagnosis that predict a more severe disease course, which would suggest the need for DMT initiation. For DMT escalation, we will evaluate the disease course of each patient over the first 3 years of follow up, using recent guidance on clinical and radiological features that suggest escalation to treatment or more effective treatment is required. These factors will be included as weighted variables to generate a summary number (0-1), the Propensity Score (PS): a higher propensity score would suggest a higher likelihood of being in the treated or escalated group.

Once each patient has been assigned a propensity score, we will assess the actual use of DMTs, matching treated and non-treated, and escalated and non-escalated patients into pairs for comparison of outcome. We anticipate that more patients with a high propensity score (and therefore a higher propensity to treatment) will have been initiated or escalated onto DMTs in Greater Glasgow in comparison to Grampian. Prognostically similar patients managed differently within a centre will also be matched, since the purpose is to compare patients and not centres. If data from the Glasgow and Grampian Centres do not provide enough propensity-matched pairs, data from the Edinburgh and Dundee centres can also be extracted.

Phase 1 - completed This retrospective phase has been completed and examined whether patients with RRMS are treated differently within Scotland despite similar disease severity. We established the proportion of patients from each centre with a high propensity score for DMT initiation or escalation who were 'treated' and 'escalated', or not, respectively. This allowed us to identify pairs for comparison of outcomes in the prospective phase of the study (Phases 2).

Phase 2 - proposed Propensity score-matched patients who were managed differently during phase 1 will be invited for a clinical assessment and MRI in the prospective phase of the study. This will be 10 years on from date of diagnosis. Contemporary clinical assessment will include physical and cognitive evaluations as detailed below. Updated radiological assessment with MRI will assess T2 and T1 lesions and total brain volume. Patients will also be asked to provide a variety of patient reported outcome measures (PROMs) by completing validated questionnaires to describe their perceived disease status. After assessments are complete, a clinical history via a structured questionnaire will be performed to capture disease activity and changing/escalation of treatment from diagnosis to point of assessment 10 years later.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Relapsing-Remitting Multiple Sclerosis (RRMS) in 2010-11 in Scotland, as held on the Scottish Multiple Sclerosis Register

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As above, Patients diagnosed with Relapsing-Remitting Multiple Sclerosis (RRMS) in 2010-11 in Scotland, as held on the Scottish Multiple Sclerosis Register
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Mean Expanded Disability Status Scale (EDSS) score at prospective assessment. | Single visit assessment competed by Dec 2022
  EDSS scores range from 0-10. The higher the score the worse the level of disability.

SECONDARY OUTCOMES:
Proportion experiencing (serious) adverse events in first 9-10 years after diagnosis | Single visit assessment competed by Dec 2022
  Proportion experiencing (serious) adverse events in first 9-10 years after diagnosis
Proportion attaining Expanded Disability Status Scale (EDSS) 3.0, 4.0 and 6.0 | Single visit assessment competed by Dec 2022
  EDSS scores range from 0-10. The higher the score the worse the level of disability.
Mean change in Expanded Disability Status Scale (EDSS) between treatment groups | Single visit assessment competed by Dec 2022
  We will be using estimated EDSS at diagnosis and actual EDSS at the prospective assessment. EDSS scores from 0-10. The higher the score the worse the level of disability.
Mean scores on patient reported outcome measure Multiple Sclerosis Impact Scale -29 (MSIS-29) at prospective assessment | Single visit assessment competed by Dec 2022
  Multiple Sclerosis Impact Scale -29 scores range from 29 to 145. The higher the score the worse the outcome
Mean Brief International Cognitive Assessment for MS (BICAMS) score at prospective assessment | Single visit assessment competed by Dec 2022
  The higher the score the better the outcome
Mean 9-Hole Peg Test (9-HPT) at prospective assessment | Single visit assessment competed by Dec 2022
  Patients are timed how long it takes to place 9 pegs into holes and then remove them, placing them in a small container. The outcome is measured in time, the quicker the time, the better the outcome

OTHER OUTCOMES:
Mean scores on patient reported outcome measures (PROMs) | Single visit assessment competed by Dec 2022
  We will ask patients to report how they view their upper and lower limb function using Neuro-quality of life score. Cognition will be assessed using Patient-Reported Outcomes Measurement Information System (PROMIS) applied cognition-abilities score. This score ranges from 41-205, the higher the score, the better the outcome
Mean volume of grey matter and whole brain volume on prospective MRI scans | Single visit assessment competed by Dec 2022
  Mean volume of grey matter and whole brain volume on prospective MRI scans
Mean lesion volume of T2/FLAIR on prospective MRI scans | Single visit assessment competed by Dec 2022
  Mean lesion volume of T2/FLAIR on prospective MRI scans

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No